CLINICAL TRIAL: NCT04879043
Title: A Phase 1/2a, First-in-human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of HDP-101 in Patients With Plasma Cell Disorders Including Multiple Myeloma
Brief Title: Study to Assess Safety of HDP-101 in Patients With Relapsed Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Heidelberg Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HDP-101-01
Record Dates: First submitted 2021-04-23; First posted 2021-05-10 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Multiple Myeloma; Plasma Cell Disorder
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Intervention Model Description: Eligible patients will be enrolled and treated with intravenous HDP-101 every 3 weeks. In Phase 1 dose-escalation part from Cohort 6 additional treatment arms are introduced for dose-optimization purposes with dosing every 3 weeks, split dosing weekly or split dosing in the first cycle on Day1 and Day8.
  A Bayesian logistic regression model will be used to guide dose-escalation during Phase 1 and select the best dose for the Phase 2a of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HDP-101 (Experimental): Participants will receive HDP-101 intravenously in a 21 day cycle until disease progression, intolerable toxicity, Investigator's discretion or patient withdrawal.
  During the phase 1 tolerability of different dose levels will be evaluated. During the phase 2a dose expansion part the recommended phase 2 dose (RP2D) of HDP-101 will be administered.
  Interventions: Drug: HDP-101

INTERVENTIONS:
Drug: HDP-101 — HDP-101 is available as lyophilized white powder for preparation of infusion.

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics (PK) and the therapeutic potential of HDP-101 in patients with plasma cell disorders including multiple myeloma.

DETAILED DESCRIPTION:
The study will consists of two parts: a Part 1 dose escalation phase and a Part 2a expansion phase for safety, tolerability, PK, PD, and clinical activity testing. The study will enroll subjects with relapsed/refractory MM or other plasma cell disorders expressing BCMA. An adaptive 2-parameter Bayesian logistic regression model (BLRM) for dose-escalation with overdose control will be used in the dose-escalation phase for determination of the MTD or the RP2D. Dose-expansion phase of the study aims to collect preliminary evidence of antitumor activity and to confirm the safety of the HDP-101 as a monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥18 years.
* Life expectancy >12 weeks.
* Eastern Cooperative Oncology Group Performance Status (PS) of 0 to 2.
* A confirmed diagnosis of active MM according to the diagnostic criteria established by the International Myeloma Working Group (IMWG).
* Must have undergone SCT or is considered transplant ineligible.
* Must have undergone prior treatments with antimyeloma therapy which must have included an immunomodulatory drug, proteasome inhibitor, and anti-CD38 treatment, alone or in combination. In addition, the patient should either refractory or intolerant to any established standard of care therapy providing a meaningful clinical benefit for the patient assessed by the Investigator.
* Measurable disease as per IMWG criteria.
* Adequate organ system function as defined in protocol.

Exclusion Criteria:

* For patient entering the Phase 2a part only: Prior treatment with any approved or experimental BCMA-targeting modalities are not allowed.
* Known central nervous system involvement.
* Plasma cell leukemia.
* History of congestive heart failure.
* Autologous or allogenic SCT within 12 weeks before the first infusion or is planning for autologous SCT.
* Symptomatic graft versus host disease post allogenic hemopoietic cell transplant within 12 months prior to the first study treatment infusion.
* Radiotherapy within 21 days prior to the first study treatment infusion.
* History of any other malignancy known to be active.
* Known human immunodeficiency virus infection.
* Patients with active infection requiring systemic anti-infective.
* Patients with positive test results for hepatitis B surface antigen or Hepatitis B core antigen.
* Patients with positive test results for hepatitis C virus (HCV) infection.
* Current active liver or biliary disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients who experience dose-limiting toxicity (DLT) during the first cycle of treatment - Part 1 as defined in Clinical Study Protocol | Up to Day 21 (from first dose)
Objective response rate (ORR) | Through study completion, an average of 1 year
  Proportion of enrolled subjects who achieve a partial response (PR) or better, i.e. stringent complete response (sCR), complete response (CR), very good partial response (VGPR) and PR, according to the IMWG criteria.

SECONDARY OUTCOMES:
Assess the safety and tolerability of HDP-101 | Through study completion, an average of 1 year
  Number of patients with serious and non-serious adverse events grouped by system organ class and preferred terms based on Common Terminology Criteria for Adverse Events (CTCAE v 5.0) classification.
To assess the anticancer activity of HDP-101 in terms of time-to-event (TTE) | Through study completion, an average of 1 year
  Clinical efficacy of HDP-101 measured by Progression Free Survival (PFS) and Overall Survival (OS).

CONTACTS AND LOCATIONS:
Locations (16):
- United States (3):
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Mount Sinai, The Tisch Cancer Instutute, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
- Germany (8):
  - Charité - Campus Benjamin Franklin Med. Klinik m.S. Hämatologie, Onkologie, Berlin
  - Klinikum Chemnitz gGmbH, Klinik f. Innere Medizin III, Chemnitz
  - Universitätsklinikum Köln, Cologne
  - Asklepios Klinik Altona, Haematologie und internistische Onkologie, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - UKSH Campus Lübeck Klinik für Hämatologie und Onkologie, Lübeck
  - Universitätsklinikum Mainz, Mainz
- Hungary (2):
  - Semmelweis University, Belgyogyaszati es Onkologiai Klinika, Budapest
  - National Institute of Oncology, Department of Oncological Internal Medicine, Budapest
- Poland (3):
  - Pratia Onkologia Katowice, Katowice
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Lodz
  - Szpital Wojewodzki w Opolu, Opole

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strassz A, Raab MS, Orlowski RZ, Kulke M, Schiedner G, Pahl A. A First in Human Study Planned to Evaluate HDP-101, an Anti-BCMA Amanitin Antibody-Drug Conjugate with a New Payload and a New Mode of Action, in Multiple Myeloma. Blood 2020; 136 (Supplement 1): 34. doi: https://doi.org/10.1182/blood-2020-142285